CLINICAL TRIAL: NCT04529525
Title: Ivermectin to Prevent Hospitalizations in COVID-19: Randomized, Double-blind, Placebo-controlled
Brief Title: Ivermectin to Prevent Hospitalizations in COVID-19
Acronym: IVERCORCOVID19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto de Cardiología de Corrientes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVERCORCOVID19MSPICC
Record Dates: First submitted 2020-08-21; First posted 2020-08-27 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2020-09

CONDITIONS: Covid19
Keywords: Ivermectin
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivermectin (Active Comparator): The dose of ivermectin in patients who are randomized to the active substance depends on the weight of the patient:
  More than 48 kg and less than 80 kg: Two tablets of 6 mg each (12 mg in total) at the time of inclusion and the same dose at 24 hours.
  More than 80 kg and less than 110 kg: Three tablets of 6 mg each (18 mg in total) at the time of inclusion and the same dose at 24 hours.
  More than 110 Kg: Four tablets of 6 mg each (24 mg in total) at the time of inclusion and the same dose at 24 hours.
  Interventions: Drug: Ivermectin
- Placebo (Placebo Comparator): The dose of placebo in patients who are randomized to the this depends on the weight of the patient:
  More than 48 kg and less than 80 kg: Two tablets of 6 mg each (12 mg in total) at the time of inclusion and the same dose at 24 hours.
  More than 80 kg and less than 110 kg: Three tablets of 6 mg each (18 mg in total) at the time of inclusion and the same dose at 24 hours.
  More than 110 Kg: Four tablets of 6 mg each (24 mg in total) at the time of inclusion and the same dose at 24 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivermectin — Patients will receive the tablet from the branch to which they were randomized only at the time of inclusion and 24 hours after the first dose.
  Arms: Ivermectin
Drug: Placebo — Patients will receive the tablet from the branch to which they were randomized only at the time of inclusion and 24 hours after the first dose.
  Arms: Placebo

SUMMARY:
It is a single-center, prospective, randomized, double-blind, placebo-controlled study carried out by the Ministry of Public Health of the Province of Corrientes, Argentina, in coordination with the Corrientes Institute of Cardiology "Juana F. Cabral". Patients who meet all the inclusion criteria and none of the exclusion criteria are randomized via the web system to receive placebo or ivermectin. The need for hospitalization in patients with COVID-19 is assessed as the primary end point. As secondary end points are evaluated: time to hospitalization (in days); use of invasive mechanical ventilation; time to invasive mechanical ventilation (in days); dialysis; all-cause mortality; negative of the swab at 3 ± 1 days and 12 ± 2 days after entering the study and ivermectin safety.

Intermediate internal analyzes of study objectives and serious adverse events will be performed, including 125; 250 and 375 patients in order to assess the possible need for early termination of the study. For these intermediate internal analyzes, the Haybittle-Peto rule will be followed, therefore a value of p <0.001 will be considered significant

DETAILED DESCRIPTION:
The study will be carried out in the province of Corrientes, in the Argentine Republic. All patients must be domiciled in this province. In the province of Corrientes, the care of patients with COVID19 is in charge of a single group of professionals (Crisis Committee) and patients who require hospitalization will be carried out in a single hospital destined for this purpose

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age who reside in the province of Corrientes at the time of diagnosis;
* Confirmed diagnosis of COVID-19 by polymerase chain reaction test for detection of SARS-CoV2 in the last 48 hours;
* In the case of women of childbearing age, they must be using a contraceptive method of proven efficacy and safety (barrier, hormonal or permanent contraceptives) for at least 3 months prior to inclusion in the present study and for the entire period of time for the duration of the study and until at least 30 days after the end of this study. A woman will be considered to have no reproductive capacity if she is postmenopausal (at least 2 years without her menstrual cycles) or if she has undergone surgical sterilization (at least one month before the time of inviting her to participate in this study);
* Weight at the time of inclusion greater than 48,000 kilograms;
* That they sign the informed consent for participation in the study.

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Known allergy to ivermectin or some of the components of ivermectin tablets or placebo;
* Current use of home oxygen;
* That require hospitalization due to COVID-19 at the time of diagnosis or history of hospitalization for COVID-19;
* Presence of mal-absorptive syndrome;
* Presence of any other concomitant acute infectious disease;
* Known history of severe liver disease, for example liver cirrhosis;
* Need or use of antiviral drugs at the time of admission for another viral pathology other than COVID-19;
* Need or use of hydroxychloroquine or chloroquine;
* Use of ivermectin up to 7 days prior to randomization;
* Patients on dialysis or who have required it in the last 2 months or who plan to do it in the next 2 months;
* Current participation or in the last 30 days in a research study that has included the administration of a drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
Percentage of Hospitalization of medical cause in patients with COVID-19 in each arm | through study completion, an average of 30 days
  Hospitalization will be considered when at least 24 hours have elapsed in a health institution, in any of its services.

SECONDARY OUTCOMES:
Time to hospitalization | through study completion, an average of 30 days
  Number of days elapsed
Percentage of Use of invasive mechanical ventilation support in each arm | through study completion, an average of 30 days
  All patients who are connected to invasive mechanical ventilation support
Time to invasive mechanical ventilation support | through study completion, an average of 30 days
  Number of days elapsed
Percentage of dialysis in each arm | through study completion, an average of 30 days
  All patients who require temporary or permanent renal replacement therapy
All-cause mortality | through study completion, an average of 30 days
  Death of the patient, from any cause.
Negative of the swab at 3±1 days and 12±2 days after entering the study | At days 3±1 and 12±2
  Negative Nasal Swab Using Polymerase Chain Reaction Technique
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | through study completion, an average of 30 days
  According to the adverse events that patients may present.

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Public Health of the Province of Corrientes, Corrientes, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Simsek Yavuz S, Unal S. Antiviral treatment of COVID-19. Turk J Med Sci. 2020 Apr 21;50(SI-1):611-619. doi: 10.3906/sag-2004-145. PMID 32293834
- [Result] Gonzalez Canga A, Sahagun Prieto AM, Diez Liebana MJ, Fernandez Martinez N, Sierra Vega M, Garcia Vieitez JJ. The pharmacokinetics and interactions of ivermectin in humans--a mini-review. AAPS J. 2008;10(1):42-6. doi: 10.1208/s12248-007-9000-9. Epub 2008 Jan 25. PMID 18446504
- [Result] Gotz V, Magar L, Dornfeld D, Giese S, Pohlmann A, Hoper D, Kong BW, Jans DA, Beer M, Haller O, Schwemmle M. Influenza A viruses escape from MxA restriction at the expense of efficient nuclear vRNP import. Sci Rep. 2016 Mar 18;6:23138. doi: 10.1038/srep23138. PMID 26988202
- [Result] Lundberg L, Pinkham C, Baer A, Amaya M, Narayanan A, Wagstaff KM, Jans DA, Kehn-Hall K. Nuclear import and export inhibitors alter capsid protein distribution in mammalian cells and reduce Venezuelan Equine Encephalitis Virus replication. Antiviral Res. 2013 Dec;100(3):662-72. doi: 10.1016/j.antiviral.2013.10.004. Epub 2013 Oct 22. PMID 24161512
- [Result] Tay MY, Fraser JE, Chan WK, Moreland NJ, Rathore AP, Wang C, Vasudevan SG, Jans DA. Nuclear localization of dengue virus (DENV) 1-4 non-structural protein 5; protection against all 4 DENV serotypes by the inhibitor Ivermectin. Antiviral Res. 2013 Sep;99(3):301-6. doi: 10.1016/j.antiviral.2013.06.002. Epub 2013 Jun 14. PMID 23769930
- [Result] Wagstaff KM, Sivakumaran H, Heaton SM, Harrich D, Jans DA. Ivermectin is a specific inhibitor of importin alpha/beta-mediated nuclear import able to inhibit replication of HIV-1 and dengue virus. Biochem J. 2012 May 1;443(3):851-6. doi: 10.1042/BJ20120150. PMID 22417684
- [Result] Chi NC, Adam EJ, Adam SA. Sequence and characterization of cytoplasmic nuclear protein import factor p97. J Cell Biol. 1995 Jul;130(2):265-74. doi: 10.1083/jcb.130.2.265. PMID 7615630
- [Result] Gorlich D, Mattaj IW. Nucleocytoplasmic transport. Science. 1996 Mar 15;271(5255):1513-8. doi: 10.1126/science.271.5255.1513. PMID 8599106
- [Result] Rowland RR, Chauhan V, Fang Y, Pekosz A, Kerrigan M, Burton MD. Intracellular localization of the severe acute respiratory syndrome coronavirus nucleocapsid protein: absence of nucleolar accumulation during infection and after expression as a recombinant protein in vero cells. J Virol. 2005 Sep;79(17):11507-12. doi: 10.1128/JVI.79.17.11507-11512.2005. PMID 16103202
- [Result] Timani KA, Liao Q, Ye L, Zeng Y, Liu J, Zheng Y, Ye L, Yang X, Lingbao K, Gao J, Zhu Y. Nuclear/nucleolar localization properties of C-terminal nucleocapsid protein of SARS coronavirus. Virus Res. 2005 Dec;114(1-2):23-34. doi: 10.1016/j.virusres.2005.05.007. Epub 2005 Jun 29. PMID 15992957
- [Result] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768
- [Derived] Vallejos J, Zoni R, Bangher M, Villamandos S, Bobadilla A, Plano F, Campias C, Chaparro Campias E, Medina MF, Achinelli F, Guglielmone HA, Ojeda J, Farizano Salazar D, Andino G, Kawerin P, Dellamea S, Aquino AC, Flores V, Martemucci CN, Martinez SM, Segovia JE, Reynoso PI, Sosa NC, Robledo ME, Guarrochena JM, Vernengo MM, Ruiz Diaz N, Meza E, Aguirre MG. Ivermectin to prevent hospitalizations in patients with COVID-19 (IVERCOR-COVID19) a randomized, double-blind, placebo-controlled trial. BMC Infect Dis. 2021 Jul 2;21(1):635. doi: 10.1186/s12879-021-06348-5. PMID 34215210
- [Derived] Vallejos J, Zoni R, Bangher M, Villamandos S, Bobadilla A, Plano F, Campias C, Chaparro Campias E, Achinelli F, Guglielmone HA, Ojeda J, Medina F, Farizano Salazar D, Andino G, Ruiz Diaz NE, Kawerin P, Meza E, Dellamea S, Aquino A, Flores V, Martemucci CN, Vernengo MM, Martinez SM, Segovia JE, Aguirre MG. Ivermectin to prevent hospitalizations in patients with COVID-19 (IVERCOR-COVID19): a structured summary of a study protocol for a randomized controlled trial. Trials. 2020 Nov 24;21(1):965. doi: 10.1186/s13063-020-04813-1. PMID 33234158